CLINICAL TRIAL: NCT01139372
Title: An Evaluation of the Daytime Use of an Investigational Lubricant Eye Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-10-006
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: Dry eye, artificial tears
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 115958D (Experimental): Lubricant eye drop
  Interventions: Other: FID 115958D (Lubricant Eye Drop)

INTERVENTIONS:
Other: FID 115958D (Lubricant Eye Drop) — 1 drop in each eye at least twice daily

SUMMARY:
The purpose of this study is to describe the subjective assessments of an investigational lubricant eye drop.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of dry eye
* Current use of Refresh Liquigel, GenTeal Gel Drops or Refresh Celluvisc at least twice daily

Exclusion Criteria:

* Must not have worn contact lenses within 7 days preceding enrollment
* Must not have had punctal plugs inserted within 30 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Daytime Use Assessment: "I would use this product at bedtime for my dry eye symptoms" Likert scale (i.e. strongly disagree, disagree, neither disagree nor agree, agree, strongly agree) | Day 7